CLINICAL TRIAL: NCT03771534
Title: Transposition of the Great Arteries: Prenatal Anatomical and Hemodynamic Findings Associated With Perinatal Outcomes
Brief Title: Acute Maternal Hyperoxygenation for Fetal Transposition of the Great Arteries (TGA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Edgar Jaeggi, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000060514
Record Dates: First submitted 2018-10-11; First posted 2018-12-11 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: TGA - Transposition of Great Arteries
Keywords: maternal hyperoxygenation; fetal echocardiography; fetal MRI
MeSH Terms: conditions — Transposition of Great Vessels | interventions — nitrox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxygen gas (Experimental): 10-15 L/min of oxygen by face mask for up to 45 minutes for the MRI and up to 30 minutes for the echocardiogram.
  Interventions: Drug: Oxygen gas

INTERVENTIONS:
Drug: Oxygen gas — Brief maternal administration of 65-70% O2 via a face mask during the last trimester
  Other Names: Praxair

SUMMARY:
This prospective study will examine whether transient maternal hyperoxygenation is useful as a diagnostic test to more accurately detect TGA patients with poor vs. good neonatal intra-cardiac mixing of blood, based on the in-utero response to oxygen exposure. This study is Health Canada regulated

DETAILED DESCRIPTION:
This is a prospective pilot study to examine whether transient maternal hyperoxygenation is useful as a diagnostic test to more accurately detect TGA patients with poor vs. good neonatal intracardiac mixing of blood, based on the in-utero response to oxygen exposure. Acute maternal oxygen administration will transiently increase the fetal oxygen levels to those reached at birth with spontaneous breathing, thus simulating conditions that will naturally occur at the time of birth. Echocardiogram and MRI will be used to examine the effects on the fetal circulation. The prenatal findings will then be compared to the neonatal presentation.

The investigators postulate that conditions that predispose newborns to acute neonatal compromise will be detectable and distinguishable prior to birth by echocardiography, MRI, or by combining the findings of both exams.

ELIGIBILITY:
Inclusion Criteria:

* Fetus with simple TGA +/- small VSD
* Intention of active postnatal management after birth

Exclusion Criteria:

* Fetus with complex form of TGA
* Significant fetal arrhythmia
* Major non-cardiac lesions
* Maternal contraindications for fetal MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Fetal intracardiac/ductal shunting measured by echocardiogram flow patterns and MRI fluximetry | Outcome measure obtained during hyperoxygenation while undergoing echocardiography and MRI
  Characterize effects of maternal hyperoxygenation on fetal intracardiac shunting measured using MRI fluximetry (ml/min/m2) of AAo, DA, SVC, IVC, UV, and DA.
  Ductal shunting measured using echo measurements of atrial septal morphology (2D; 4D) and foramen flow (color; 4D flow) of FO diameter and septal excursion. Ductus arteriosus flow (color and Doppler): minimal diameter, reversed end-diastolic flow, systolic peak flow, forward-reverse flow ratio, flow restriction.
Fetal pulmonary blood flow measured by MRI fluximetry | Outcome measure obtained during hyperoxygenation while undergoing echocardiography and MRI
  Characterize effects of maternal hyperoxygenation on fetal pulmonary blood flow using MRI fluximetry (ml/min/m2) measures of Main PA, RPA and LPA
Neonatal outcomes | Intrauterine demise to hospital discharge, or up to 1 year of age if pulmonary hypertension exists
  As measure of patient morbidity, a composite score of 10 variables will be used, assigning a value of 1 for each event that occurred 1) respiratory distress syndrome requiring surfactant; 2) cardiopulmonary resuscitation requiring chest compressions; 3) cerebral vascular injury (intra-ventricular or -parenchymal hemorrhage, ischemic stroke); 4) necrotizing enterocolitis; 5) need of ECMO; 6) infections associated with health care (bloodstream, surgical site, and urinary tract infection); 7) unplanned re-intubation; 8) re-operation for residual cardiac lesions; 9) interventional catheterization for residual cardiac lesions; and 10) unplanned intensive care readmission.

SECONDARY OUTCOMES:
Fetal cerebral perfusion | Outcome measure obtained during maternal hyperoxygenation while undergoing echocardiography and MRI
  Effects of maternal hyperoxygenation on fetal cerebral perfusion measured by change in cDO2 (mL/min/m2) and cVO2 (mL/min/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Jaeggi, MD, Principal Investigator — The Hospital for Sick Children, Toronto; Mike Seed, MBBS, Principal Investigator — The Hospital for Sick Children, Toronto
Locations (1):
- The Hospital For Sick Children, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun L, Macgowan CK, Portnoy S, Sled JG, Yoo SJ, Grosse-Wortmann L, Jaeggi E, Kingdom J, Seed M. New advances in fetal cardiovascular magnetic resonance imaging for quantifying the distribution of blood flow and oxygen transport: Potential applications in fetal cardiovascular disease diagnosis and therapy. Echocardiography. 2017 Dec;34(12):1799-1803. doi: 10.1111/echo.13760. PMID 29287129
- [Background] Porayette P, Madathil S, Sun L, Jaeggi E, Grosse-Wortmann L, Yoo SJ, Hickey E, Miller SP, Macgowan CK, Seed M. MRI reveals hemodynamic changes with acute maternal hyperoxygenation in human fetuses with and without congenital heart disease. Prenat Diagn. 2016 Mar;36(3):274-81. doi: 10.1002/pd.4762. Epub 2016 Feb 9. PMID 26701792
- [Background] Sun L, Macgowan CK, Sled JG, Yoo SJ, Manlhiot C, Porayette P, Grosse-Wortmann L, Jaeggi E, McCrindle BW, Kingdom J, Hickey E, Miller S, Seed M. Reduced fetal cerebral oxygen consumption is associated with smaller brain size in fetuses with congenital heart disease. Circulation. 2015 Apr 14;131(15):1313-23. doi: 10.1161/CIRCULATIONAHA.114.013051. Epub 2015 Mar 11. PMID 25762062
- [Background] Porayette P, van Amerom JF, Yoo SJ, Jaeggi E, Macgowan CK, Seed M. MRI shows limited mixing between systemic and pulmonary circulations in foetal transposition of the great arteries: a potential cause of in utero pulmonary vascular disease. Cardiol Young. 2015 Apr;25(4):737-44. doi: 10.1017/S1047951114000870. Epub 2014 Jun 16. PMID 24932863
- [Background] Prsa M, Sun L, van Amerom J, Yoo SJ, Grosse-Wortmann L, Jaeggi E, Macgowan C, Seed M. Reference ranges of blood flow in the major vessels of the normal human fetal circulation at term by phase-contrast magnetic resonance imaging. Circ Cardiovasc Imaging. 2014 Jul;7(4):663-70. doi: 10.1161/CIRCIMAGING.113.001859. Epub 2014 May 29. PMID 24874055
- [Background] Mawad W, Chaturvedi RR, Ryan G, Jaeggi E. Percutaneous Fetal Atrial Balloon Septoplasty for Simple Transposition of the Great Arteries With an Intact Atrial Septum. Can J Cardiol. 2018 Mar;34(3):342.e9-342.e11. doi: 10.1016/j.cjca.2017.12.010. Epub 2017 Dec 15. PMID 29398177
- [Background] Jaeggi E, Renaud C, Ryan G, Chaturvedi R. Intrauterine therapy for structural congenital heart disease: Contemporary results and Canadian experience. Trends Cardiovasc Med. 2016 Oct;26(7):639-46. doi: 10.1016/j.tcm.2016.04.006. Epub 2016 Apr 22. PMID 27234352

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03771534/Prot_SAP_002.pdf
  • Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT03771534/ICF_003.pdf